CLINICAL TRIAL: NCT03275571
Title: The Effects of Computerized Cognitive Behavior Therapy (cCBT) on Brain Health: A Feasibility Study
Brief Title: HIV, Computerized Depression Therapy & Cognition
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment rate, parent study has ended
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Marie-Josée Brouillette, Associate Professor, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-3508
Record Dates: First submitted 2017-09-06; First posted 2017-09-07 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: HIV Infections; Depression; CBT
Keywords: Cognition; Intervention; Therapy
MeSH Terms: conditions — HIV Infections; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cCBT intervention (Experimental): Over the course of 9 weeks, 30 min online sessions, once per week, with a fictive therapist.
  Interventions: Behavioral: cCBT intervention

INTERVENTIONS:
Behavioral: cCBT intervention — During each 30 minutes sessions, the participants will learn key concepts on depression, then will apply them to the program's main character who suffers from depression, and then will apply those techniques to their own personal challenges.

SUMMARY:
Among people with HIV, the severity of depressive symptoms has repeatedly been associated with the presence of self-reported cognitive difficulties, even in the absence of impairment on neuropsychological testing. There is uncertainty about the clinical importance of these self-reports, especially when neuropsychological testing is normal.

However, there is growing evidence that these self-reports are clinically important. For example, among patients with major depressive disorder (MDD), evidence suggests that functional impairments is mediated by self-reported cognitive dysfunction, rather than objective cognitive dysfunction. Treatment of depression with Cognitive-Behaviour Therapy (CBT) has been shown to improve depressive symptoms and psychosocial functioning in patients with recurrent major depressive disorder, but there are few studies of the impact of psychotherapy on self-reported cognition and cognitive performance. Good Days Ahead (GDA) is a computerized treatment program developed to address symptoms of depression and anxiety. It teaches the basic principles of computerized behavioral therapy (CBT) in nine therapy sessions, each typically taking 30 minutes to complete. GDA has been found to be as effective as face-to-face CBT in decreasing symptoms of depression and anxiety.

The hypothesis is that people whose depressive symptoms are reduced following treatment with cCBT will also report fewer cognitive difficulties than before treatment. A second hypothesis is that changes in self-reported cognition will be concordant with changes in cognitive performance, such that people who make no improvement in self-report cognition will also show no improvement in cognitive performance and those who do improve on self-report will improve on cognitive performance.

DETAILED DESCRIPTION:
Among people with HIV, the severity of depressive symptoms has repeatedly been associated with the presence of self-reported cognitive difficulties, even in the absence of impairment on neuropsychological testing. There is uncertainty about the clinical importance of these self-reports, especially when neuropsychological testing is normal, as they are thought to be susceptible to patients' biases and insights into their illness.

However, there is growing evidence that these self-reports are clinically important. Among patients with major depressive disorder (MDD), evidence suggests that functional impairments is mediated by self-reported cognitive dysfunction, rather than objective cognitive dysfunction. For example, Buist-Bouwman et al reported that more than one-quarter of the impact of MDD on work loss was directly attributable to self-reported cognitive difficulties and that cognition was a significant mediator of the association between MDD and work or role dysfunction.

When depression is treated with antidepressant medication, some degree of improvement on neuropsychological tests has been documented. However, many studies have evaluated cognitive outcomes before and after treatment rather than comparing them with placebo, potentially biasing the results by learning effects, which limits the strength of the conclusions that can be drawn.

Treatment of depression with Cognitive-Behaviour Therapy (CBT) has been shown to improve depressive symptoms and psychosocial functioning in patients with recurrent major depressive disorder, but there are few studies of the impact of psychotherapy on self-reported cognition and cognitive performance. In a group of patients with highly recurrent depression (≥4 episodes) over 2 years of follow-up, Conradi et al showed that those randomized to receive psycho-education plus CBT reported the presence of cognitive symptoms significantly less of the time compared to those receiving psycho-education only (15% of the time or 3.6 months compared to 47% or 11.3 months).

In the HIV population, a single study has examined the effect of treatment of depression on self-reported cognitive difficulties and performance on neuropsychological tests, as part of a randomized controlled trial of antidepressant efficacy. Following 12 weeks of antidepressant treatment, HIV+ individuals who reported a decrease in depressive symptoms also reported significantly fewer cognitive difficulties, despite an absence of improvement on neuropsychological testing.

In the context where the use of questionnaires eliciting cognitive difficulties is suggested as a first-line screening for HIV-Associated Neurocognitive Disorder, it is important to document the clinical factors that influence these self-reports in order to inform their clinical interpretation and develop interventions for individuals reporting cognitive difficulties.

Understanding and Optimizing Brain Health Now (BHN) cohort study: Cohort participants (N=840) are studied prospectively over a 27-month period with visits every 9 months. Patients complete questionnaires on mood (Hospital Anxiety Depression Scale-HADS), presence of cognitive symptoms (Patient Deficit Questionnaire-PDQ), and a computer-based evaluation of cognitive ability (B-CAM).

Computerized Cognitive-Behavioral Therapy (cCBT): A number of computerized treatment programs have been developed to address symptoms of depression and anxiety, and several meta-analyses of randomized controlled trials (RCTs) have shown evidence for their effectiveness. One such program, Good Days Ahead, teaches the basic principles of CBT in nine therapy sessions, each typically taking 30 minutes to complete. Good Days Ahead has been found to be as effective as face-to-face CBT in decreasing symptoms of depression and anxiety. Patients receiving treatment delivered by a computer can be provided with different levels of guidance and support: self-guidance, guidance by a technician who sends reminders, or guidance by a clinician. A recent meta-analysis of cCBT for depression and anxiety has shown that the treatment delivered with no guidance or support yielded, on average, a smaller effect size (Cohen's d = 0.17) than cCBT delivered with at least one hour of knowledgeable assistance during the course of therapy (Cohen's d = 0.72). Offering some assistance thus appears to be necessary for achieving better therapy outcomes.

Study Design : This study is part of a larger project based upon a cohort multiple randomized controlled design. Within a fully characterized cohort followed over time (n=840), people meeting the specific criteria for one or more interventions (here cCBT) are identified and a sample is randomly selected to receive the intervention. When the intervention is under investigation, the remaining eligible persons who do not receive the intervention serve as controls. In this study, we are not testing the effectiveness of cCBT as this has been demonstrated. Rather the researchers are focusing on changes in cognition in relation to depressive symptoms mediated by cCBT. This study is an exploration of a hypothesis using a single cohort design with two repeated measures. For exploratory studies, an N of 30 optimizes an analysis based on means under the central limit theorem.

Intervention: Participants who are eligible will receive online access to the Good Days Ahead cCBT program. Good Days Ahead is a learning module based on scientifically proven, evidence-based techniques. The program's content follows the teachings of the basic principles of CBT. The underlying platform generates customized learning experiences for each individual user with content including videos, text, quizzes and interactive exercises. The program comprises nine lessons of 30 minute each during which the user first learns the key concepts; then applies them to the program's main character who suffers from depression; and then applies those techniques to their own personal challenges (http://www.empower-interactive.com/solutions/good-days-ahead). Participants are expected to complete the nine sessions over 9-12 weeks.

As patients complete the cCBT program, their progress will be monitored by the research coordinator through a secure web site, using the program's dashboard feature that includes tracking of mood ratings, exercises, comprehension and completion rates. Participants will receive guidance during regular contacts by a trained research coordinator knowledgeable about the program and the basics of CBT.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the cohort study "Understanding and Optimizing Brain Health in HIV Now" with at least one remaining visit
* Able to communicate (understand and read) in English
* Depression subscale of the HADS (HADS-D) ≥ 8
* Presence of self-reported cognitive difficulties (PDQ) >40
* Score on the B-CAM > 14
* Willing to undergo 9 sessions of cCBT as per instructions and to have weekly contact with a research coordinator from the central site (by email or phone)
* Access to the internet

Exclusion Criteria:

• Current use of street drugs (excluding marijuana)

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
Self-reported cognitive difficulties (C3Q) | One week before the beginning of the intervention and up to 4 weeks after the end of the intervention
  The Communicating Cognitive Concerns Questionnaire evaluated cognitive concerns participants may have.

SECONDARY OUTCOMES:
Depressive symptoms measure (HADS) | One week before the beginning of the intervention and up to 4 weeks after the end of the intervention
  The Hospital Anxiety and Depression Scale is a two 7-items scale designed to rate depression and anxiety.
Cognitive Performance measure (B-CAM) | Up to 9 months before the beginning of the intervention and up to 2 months after the end of the intervention.
  The research team will be looking at changes on the B-CAM (brief cognitive ability measure)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Josee Brouillette, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Lesley Fellows, MD/DPhil, Principal Investigator — McGill University
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/71/NCT03275571/Prot_SAP_000.pdf